CLINICAL TRIAL: NCT06417359
Title: Comparison of Mesh Fixation and Non-Fixation in Laparoscopic eTEP Inguinal Hernia Repair
Brief Title: Comparison of Mesh Fixation and Non-Fixation in eTEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Eşref Ulutaş (Other)
Collaborators: Van Training and Research Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Mehmet Eşref Ulutaş, Principal Investigator, Konya City Hospital
Organization: Konya City Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65656565
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Migration of Implant; Pain; Postoperative Complications; Relapse
MeSH Terms: conditions — Pain; Postoperative Complications; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eTEP Mesh Fixation Group (Active Comparator): In 30 patients; Inguinal hernia surgery will be performed with the eTEP method and the 15x12x10 cm polyprolene patch used in this surgery will be marked with small metallic clips from the lateral, superomedial and inferomedial sides. During the surgery, the mesh will be fixed to three absorbable tacker the Cooper ligament, süpermedially and laterally. Patients whose pain scores (VAS score) are measured on the first postoperative day and who are suitable for discharge will be discharged after a pelvis x-ray is taken. One month after the surgery and 6 months later, patients will be called to the outpatient clinic and examined, their pain scores will be measured (VAS score) and pelvic radiographs will be taken. The movement of the clips marked on the patch will be compared with previous radiographs in cm.
  Interventions: Procedure: Mesh Fixation
- eTEP No Mesh Fixation Group (Experimental): In 30 patients; Inguinal hernia surgery will be performed with the eTEP method and the 15x12x10 cm polyprolene patch used in this surgery will be marked with small metallic clips from the lateral, superomedial and inferomedial sides. During the surgery, the mesh will not be fixed to the Cooper ligament. Patients whose pain scores (VAS score) are measured on the first postoperative day and who are suitable for discharge will be discharged after a pelvis x-ray is taken. One month after the surgery and 6 months later, patients will be called to the outpatient clinic and examined, their pain scores will be measured (VAS score) and pelvic radiographs will be taken. The movement of the clips marked on the patch will be compared with previous radiographs in cm.
  Interventions: Procedure: No Mesh Fixation

INTERVENTIONS:
Procedure: Mesh Fixation — That mesh will be fixation with three tackers.
  Arms: eTEP Mesh Fixation Group
Procedure: No Mesh Fixation — That mesh will not be fixation
  Arms: eTEP No Mesh Fixation Group

SUMMARY:
Inguinal hernia surgery is one of the most frequently performed procedures among general surgery cases. As with many open surgical methods, this repair is also performed laparoscopically. Among these closed methods, the one method is laparoscopic extended total extraperitoneal repair (eTEP). The benefits of laparoscope include less postoperative pain and complications, faster recovery, reduced chronic pain, and recurrence rate.

One of the recent debates regarding the laparoscopic technique is mesh fixation. Fixation of the mesh to the cooper ligament can prevent mesh migration and consequently reduce the recurrence rate. However, it has been reported that this fixation may increase postoperative pain. Several studies have reported that recurrence may be due to inadequate mesh fixation technique. In contrast, other prospective randomized studies have found relapse unrelated to mesh fixation.

In the eTEP technique, dissection is performed in a larger area than in TEP. For this reason, it can be thought that the possibility of mesh displacement is higher in the eTEP procedure. The purpose of this study is to confirm this idea with a prospective study. There are studies in the literature on mesh fixation related to the total extraperitoneal repair (TEP) technique. However, there is no study on mesh detection in the eTEP technique. The aim of the study is to compare patients who underwent withmesh fixation and without mesh fixation laparoscopic eTEP repair in terms of clinical data such as mesh displacement and hernia recurrence, chronic pain, length of hospital stay, and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral inguinal hernias,
* Patients aged 18-65.

Exclusion Criteria:

* Younger than 18 years, and older than 65 years,
* Incarcerated or strangulated inguinal hernias,
* Patients with bilateral inguinal hernias,
* Patients who are contraindicated to receive general anesthesia,
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-10-04 (Estimated)

PRIMARY OUTCOMES:
Status of Mesh Displacement | postoperative 24 hours, 1 and 6 months
  Patients who are suitable for discharge will be discharged after a pelvis x-ray is taken. One month after the surgery and 6 months later, patients will be called to the outpatient clinic and examined and pelvic radiographs will be taken. The movement of the clips marked on the patch will be compared with previous radiographs in cm.

SECONDARY OUTCOMES:
Rate of Postoperative pain | postoperative 24 hours
  It will be measured using the Visual Analog Score (VAS). The patient will be asked to choose between the number 1 with the least pain and the number 10 with the most pain. The lowest score on this scale is 1, and the highest score is 10.
Rate of Hernia recurrence | postoperative 6th month and first year
  hernia recurrence after six months of follow-up. It will be checked by physical examination. Imaging methods will be used in suspicious cases.
Rate of Postoperative complications | postoperative 24 hours and 1st month
  such as wound infection, bleeding
Rate of Chronic pain | postoperative 1st, 6th month and first year
  It will be measured using the Visual Analog Score (VAS). The patient will be asked to choose between the number 1 with the least pain and the number 10 with the most pain. The lowest score on this scale is 1, and the highest score is 10.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science Van Training and Research Hospital, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yildirim MB, Sahiner IT. The effect of mesh fixation on migration and postoperative pain in laparoscopic TEP repair: prospective randomized double-blinded controlled study. Hernia. 2023 Feb;27(1):63-70. doi: 10.1007/s10029-022-02587-w. Epub 2022 Mar 14. PMID 35286511
- [Result] Claus CMP, Rocha GM, Campos ACL, Paulin JAN, Coelho JCU. Mesh Displacement After Bilateral Inguinal Hernia Repair With No Fixation. JSLS. 2017 Jul-Sep;21(3):e2017.00033. doi: 10.4293/JSLS.2017.00033. PMID 28904521
- [Result] Claus CM, Rocha GM, Campos AC, Bonin EA, Dimbarre D, Loureiro MP, Coelho JC. Prospective, randomized and controlled study of mesh displacement after laparoscopic inguinal repair: fixation versus no fixation of mesh. Surg Endosc. 2016 Mar;30(3):1134-40. doi: 10.1007/s00464-015-4314-7. Epub 2015 Jun 20. PMID 26092029
- [Derived] Yilmaz AH, Ulutas ME. Assessment of mesh displacement following laparoscopic enhanced view totally extraperitoneal technique: comparing mesh fixation and non-fixation in difficult inguinal hernias. Updates Surg. 2025 May 28. doi: 10.1007/s13304-025-02271-5. Online ahead of print. PMID 40434603